CLINICAL TRIAL: NCT03236012
Title: Hyperhidrosis of the Residual Limb in Patients With Amputations: Developing a Treatment Approach
Brief Title: Hyperhidrosis in Patients With Amputations-Botox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colby Hansen, Principle Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_107999; OP150030 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Hyperhidrosis
Keywords: amputation, amputations, sweating, residual limb,
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A; 2-methylcyclopentadienyl manganese tricarbonyl; Blood Cell Count; Bone Morphogenetic Proteins; Vital Capacity

STUDY DESIGN:
Intervention Model Description: For this study, subjects will be recruited from the amputee clinics held at the Salt Lake Veteran Affairs (VA) Medical Center or the University of Utah. Combined, these clinics serve approximately 500 patients and see approximately 75 new patients each year.
  We plan to recruit a total of 25 subjects to this project from the two study sites. It is expected that we will enroll equal numbers from both the University of Utah and VA Medical Center.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Botulinum Toxin Therapy (Experimental): Test the effectiveness of Botulinum Toxin therapy in subjects who fail or do not tolerate Aluminum Chloride.
  We plan to conduct an open label study of Botox, up to 400 units, in amputees who have failed treatment with a topical antiperspirant.
  Interventions: Drug: Botulinum Toxin Type A (Botox)

INTERVENTIONS:
Drug: Botulinum Toxin Type A (Botox) — Maximum dose up to 400 units given one time
  Other Names: Manual Muscle Testing (MMT), Labs (CBC, BMP, PFT'S, (FEV1 & FVC)), Iodine Starch Skin Test

SUMMARY:
The objective is to establish and evidence base for hyperhidrosis treatment algorithm in amputees.This project will address a problem that has troubled Service members, Veterans, and civilians with amputations for decades, impacting satisfaction with prosthetic use, residual limb skin health, and negatively affecting quality of life. Prior research in this area has been limited and insufficient. We plan to conduct an open label study of Botox, up to 400 units, to treat limb hyperhidrosis in patients with amputations. The actual dose of Botox used will be based on individual results with the Iodine-Starch test to identify areas on the residual limb that are producing excessive sweat. Botulinum Toxin A (BTX-A): Botulinum toxin therapy is well-established for use in excessive sweating of several body areas (axillary, palmar, plantar, and facial) in individuals with hyperhidrosis and inadequate response to topical treatments. Extensive research has been conducted on the efficacy and safety of BTX-A for hyperhidrosis of other areas, and it has been shown to improve both objective and subjective measures of sweating, and lead to improved quality of life measures.

This will be accomplished by completing the following:

Test the validity of the Minor iodine-starch test in amputees.

1. Hypothesis: The iodine-starch test is a valid diagnostic tool of hyperhidrosis and can be useful for the identification of focal areas of sweating on a residual limb.
2. Treat the residual limb Hyperhidrosis with Botox, up to and limited to 400 units.

Hypothesis: Treatment of residual limb Hyperhidrosis with Botox will result in improved patient reports of excessive sweating as measured by the HDSS and as measured by subjects' response to iodine-starch testing. We are confident that improving the evaluation and treatment of residual limb hyperhidrosis will reduce the secondary health consequences of amputation and will lead to improved quality of life.

DETAILED DESCRIPTION:
Subjects who meet inclusion criteria will be given Botox injections. The maximum dose that will be used will vary from patient to patient up to 400 units.

We will test the effectiveness of botulinum toxin therapy in those who fail Aluminum Chloride. Failure will be defined as a non-response (no change in HDSS), inadequate response (post-treatment HDSS of 2 or more), or intolerance to Aluminum Chloride. This would be a natural progression of interventions consistent with guidelines for other forms of hyperhidrosis. Specifically, we will study botulinum toxin type A BTX-A, brand name Botox. While there are other BTX-A products on the market, Botox is the only FDA approved toxin for the treatment of axillary hyperhidrosis.

There are a few considerations to make when dosing Botox for hyperhidrosis. These include the total dose, the dose per injection site, and the distribution of injection sites. Typical doses for axillary hyperhidrosis are 50- 100 units per axilla18. However, for clinical trials used to support the FDA-approved labeling in focal spasticity, doses up to 400 units were used. There are reports of off label dosing exceeding this amount, including the case series reported by Charrow for residual limb hyperhidrosis, which used doses ranging from 300 - 500 units of Botox. There was no mention of adverse events in this series. It has been suggested that doses greater than 600 units pose a greater risk of serious adverse events including systemic weakness. Regarding dose per injection site, hyperhidrosis guidelines suggest 1 unit per site for the axilla, and 1.5 - 2 units per site for the palm or sole18. The largest case series in amputees used doses of 2-3 units per site. Regarding the distribution of injection sites, guidelines recommend injections every 1 - 2 cm in a grid-like fashion.

We plan to conduct an open label study of Botox, up to 400 units, in amputees who have failed treatment with a topical antiperspirant.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated informed consent form (ICF)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, age 18 or older
* At least 6 months post-amputation surgery
* Have a prosthetic device
* In good general health as evidenced by medical history
* HDSS score of 2 or greater AND failed prior treatment with topical Aluminum Chloride.
* At least 6 months from last injection with any botulinum toxin

Exclusion Criteria

* Open sores or wounds on the residual limb
* Known sensitivity or allergy to iodine
* Pregnancy or lactation
* Any prior Hypersensitivity reaction to Botox including anaphylaxis, serum sickness, urticaria, soft tissue edema, and dyspnea
* Infection at the injection site
* Known neuromuscular junction disorder
* Inflammation at the injection site
* A known compromised respiratory status which may include the use of oxygen, recent hospitalization for respiratory illness, including but not limited to recent antibiotic treatment for pneumonia, bronchitis or other respiratory tract infections will not be allowed to participate
* Overactive bladder with a history of recurrent urinary tract infection (UTI) or two or more UTI's

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
The effectiveness of botulinum toxin therapy in subjects who fail Aluminum Chloride as assessed by the Hyperhidrosis Disease Severity Scale (HDSS) | Baseline to 20 weeks
  The outcome measure for this study will be measuring the Hyperhidrosis Disease Severity Scale (HDSS). The HDSS is scored on a number scale of 1-4. Score range from 1 (lowest) demonstrating sweating (hyperhidrosis) is least noticeable and does not interfere with daily activities (least impactful) to 4 (highest) sweating is intolerable and interferes significantly with daily activities. This measurement will be completed at Baseline, Week #4 clinic visit, Week #12 clinic visit, Week#16 clinic visit and week#20 follow up phone call visit.

SECONDARY OUTCOMES:
The effectiveness of botulinum toxin therapy in subjects who fail Aluminum Chloride as assessed by the Sweating Intensity Visual Scale (SIVS) | Baseline to 20 weeks
  The secondary outcome measure for this study will be measuring the Sweating Intensity Visual Scale (SIVS). The SIVS is assessed on a number scale of 0-5. A score of zero (lowest) indicates no effect from sweating (hyperhidrosis) relating to the fit and functioning of the prosthesis (least impactful) to 5 (highest) which means severely affecting the fit and functioning of the prosthesis. This measurement will be completed at Baseline, Week# 4 clinic visit, Week #12 clinic visit, Week#16 clinic visit and week#20 follow up phone call visit.

CONTACTS AND LOCATIONS:
Overall Officials: Colby Hansen, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah Hospital, Salt Lake City, Utah
  - George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided